CLINICAL TRIAL: NCT03508297
Title: Reflectance Confocal Microscopy to Diagnose Malignant Melanoma and Lentigo Maligna
Brief Title: Reflectance Confocal Microscopy to Diagnose MM & LM
Status: Completed | Type: Observational
Sponsor: Skin Care Network Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HS-MAV-002
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Melanoma (Skin); Lentigo Maligna
Keywords: Confocal; RCM; Imaging; Skin cancer
MeSH Terms: conditions — Melanoma; Hutchinson's Melanotic Freckle; Skin Neoplasms | interventions — Intravital Microscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: In-vivo imaging — Skin cancer is imaged using RCM and a diagnosis is recorded before patient is returned to standard of care (biopsy).

SUMMARY:
A reflectance confocal microscope is a machine which is able to examine the upper layers of the skin painlessly and without the need for taking a biopsy. We would like to examine the images taken by the confocal microscope to see if it can help more accurately identify lesions which are worrying rather than a benign mole. We are performing this study in patients in whom we have recommended excising a mole to exclude a cancer. If the results of the study show that the confocal microscope can help more accurately diagnose Melanomas then this would reduce the number of biopsies that are taken that turn out not to be cancerous (ie unnecessary biopsies).

DETAILED DESCRIPTION:
Study Design This is an observational, non-randomised, non-controlled, prospective cohort study to look at the efficacy of in vivo RCM as a diagnostic tool in the diagnosis of MM and LM.

Study Endpoints The hypothesis of this study is that the use of RCM is would reduce the NNE prior to definitive treatment by at least 30% from the current value of approximately 10.

The secondary hypothesis is that the intra- & inter-observer agreement for interpreting the RCM images will have kappa scores 0.6 or greater (indicating good agreement).

Setting and recruitment Patients will be recruited from the outpatient clinics of the Skin Care Network Barnet, and from the outpatient clinics of the Chase Farm and Barnet sites of Royal Free Hospital NHS Foundation Trust.

Participants The number of true negative lesions examined in this study will be 654. It is anticipated that this will result in a total of 661 lesions being recruited. 10% of participants are expected to have more than one lesion sampled.

The result of biopsy for each lesion will not be known until after the lesion has been included in the study. Therefore lesions will be added to the study until the required number of true negatives has been included.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Patient with a pigmented lesion recommended for excision because of suspicion of MM or LM.
3. Patient willing and able to give informed consent

Exclusion Criteria:

1. Recurrent MM or LM
2. Patient on immunosuppresants
3. Patient with significant co-morbidity or skin disease
4. Patient not suitable for diagnostic biopsy
5. Location of lesion unsuitable, inaccessible or impractical for scanning with RCM as determined by investigator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients presenting at a skin cancer clinic with a lesion that is clinically suspicious for LM or MM.
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Number Needed to Excise | During exam (biopsy results typically available within one week).
  The number of suspicious lesions (defined by conventional histology) biopsied to find one cancerous lesion

SECONDARY OUTCOMES:
intra- & inter-observer agreement for interpreting the RCM images will have kappa scores 0.6 or greater | 6 months
  A measure of how consistently readers can diagnose from confocal images.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Stevens, MA PhD, Principal Investigator — Skin Care Network Ltd.
Locations (1):
- Skin Care Network Barnet Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stevens HP, Pellacani G, Angus C, El-Jabbour JN. Reflectance confocal microscopy to diagnose malignant melanoma and lentigo maligna in the UK: a single-centre prospective observational trial. Br J Dermatol. 2024 Dec 23;192(1):27-35. doi: 10.1093/bjd/ljae354. PMID 39255055

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT03508297/Prot_SAP_000.pdf